CLINICAL TRIAL: NCT00106158
Title: Immunization of Patients With Tumors Expressing NY-ESO-1 or LAGE Antigen With Complex of NY-ESO-1 Protein and Cholesterol-bearing Hydrophobized Pullulan (CHP)
Brief Title: Safety Study of NY-ESO-1 Protein Vaccine to Treat Cancer Expressing NY-ESO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2002-005
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2007-08

CONDITIONS: Neoplasms
Keywords: cancer/testis antigen; cancer vaccine; recombinant protein
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Biological: protein vaccination

SUMMARY:
The purpose of this study is to assess the safety of repeated doses of cholesterol-bearing hydrophobized pullulan (CHP) and NY-ESO-1 protein (CHP-NY-ESO-1) and describe the NY-ESO-1 specific-humoral and cellular immune response to immunization with CHP-NY-ESO-1 in patients with cancer expressing NY-ESO-1.

DETAILED DESCRIPTION:
NY-ESO-1 was isolated by serological analysis of recombinant cDNA expression libraries (SEREX), using tumor mRNA and autologous serum from an esophageal cancer patient. Reverse transcription-polymerase chain reaction (RT-PCR) analysis showed that NY-ESO-1 displayed the typical expression pattern of CT antigens. NY-ESO-1 mRNA was expressed only in testis of normal tissues tested and in various types of cancer, including lung cancer, breast cancer, malignant melanoma and bladder cancer. LAGE-1 was identified by the representational difference analysis and revealed to display 84% amino acid homology with NY-ESO-1. In most cases, expression of LAGE-1 parallels the expression of NY-ESO-1. Since testis is an immune privileged organ where HLA molecules are not expressed, these antigens can be considered tumor-specific.

Because of frequent NY-ESO-1 mRNA expression and high immunogenicity in advanced cancer, NY-ESO-1 is an attractive target molecule for a cancer vaccine. Current therapies against advanced cancer have limited effectiveness. The idea of vaccination with NY-ESO-1 protein in cancer patients with tumors expressing NY-ESO-1 mRNA is based on two findings: 1) the number of CD8+ T cell epitopes identified in NY-ESO-1 molecule are limited to those binding to HLA-A0201, A31, Cw3 and Cw6. These HLA subtypes are carried by a minor Japanese population; 2) CD8+ T cell responses specific to NY-ESO-1 are polyclonal. Protein vaccination may induce immune response more effectively against tumors expressing NY-ESO-1 than peptide immunization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven cancer
* Confirmed NY-ESO-1 expression
* No other effective therapy available
* 4 weeks since conventional therapy before start of the current protocol
* Performance status < 2 (ECOG scale)
* Age > 18
* Able and willing to give written informed consent

Exclusion Criteria:

* Serious illness
* Metastatic diseases to central nervous system
* Concomitant systemic treatment with corticosteroids, anti-histaminic drugs or NSAIDs
* HIV positive
* Mental impairment that may compromise the ability to give written informed consent
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2004-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
NY-ESO-1-specific immune responses

SECONDARY OUTCOMES:
tumor responses

CONTACTS AND LOCATIONS:
Overall Officials: Eiichi Nakayama, MD., PhD, Principal Investigator — Dept. of Immunology, Okayama University Schhol of Medicine and Dentistry
Locations (1):
- Dept. of Immunology, Okayama University School of Medicine and Dentistry, Okayama, Japan

REFERENCES:
- [Background] Sato S, Noguchi Y, Wada H, Fujita S, Nakamura S, Tanaka R, Nakada T, Hasegawa K, Nakagawa K, Koizumi F, Ono T, Nouso K, Jungbluth A, Chen YT, Old LJ, Shiratori Y, Nakayama E. Quantitative real-time RT-PCR analysis of NY-ESO-1 and LAGE-1a mRNA expression in normal tissues and tumors, and correlation of the protein expression with the mRNA copy number. Int J Oncol. 2005 Jan;26(1):57-63. PMID 15586225
- [Background] Sugita Y, Wada H, Fujita S, Nakata T, Sato S, Noguchi Y, Jungbluth AA, Yamaguchi M, Chen YT, Stockert E, Gnjatic S, Williamson B, Scanlan MJ, Ono T, Sakita I, Yasui M, Miyoshi Y, Tamaki Y, Matsuura N, Noguchi S, Old LJ, Nakayama E, Monden M. NY-ESO-1 expression and immunogenicity in malignant and benign breast tumors. Cancer Res. 2004 Mar 15;64(6):2199-204. doi: 10.1158/0008-5472.can-03-3070. PMID 15026363
- [Background] Nakada T, Noguchi Y, Satoh S, Ono T, Saika T, Kurashige T, Gnjatic S, Ritter G, Chen YT, Stockert E, Nasu Y, Tsushima T, Kumon H, Old LJ, Nakayama E. NY-ESO-1 mRNA expression and immunogenicity in advanced prostate cancer. Cancer Immun. 2003 Jul 31;3:10. PMID 12889868
- [Background] Fujita S, Wada H, Jungbluth AA, Sato S, Nakata T, Noguchi Y, Doki Y, Yasui M, Sugita Y, Yasuda T, Yano M, Ono T, Chen YT, Higashiyama M, Gnjatic S, Old LJ, Nakayama E, Monden M. NY-ESO-1 expression and immunogenicity in esophageal cancer. Clin Cancer Res. 2004 Oct 1;10(19):6551-8. doi: 10.1158/1078-0432.CCR-04-0819. PMID 15475443
- [Background] Kurashige T, Noguchi Y, Saika T, Ono T, Nagata Y, Jungbluth A, Ritter G, Chen YT, Stockert E, Tsushima T, Kumon H, Old LJ, Nakayama E. Ny-ESO-1 expression and immunogenicity associated with transitional cell carcinoma: correlation with tumor grade. Cancer Res. 2001 Jun 15;61(12):4671-4. PMID 11406534